CLINICAL TRIAL: NCT04030221
Title: The Pressure Gradient for Venous Return (PVR) in Predicting Fluid Responsiveness in Patients Undergoing Laparoscopic Surgery
Brief Title: Pressure Gradient for Venous Return in Predicting Fluid Responsiveness in Patients Undergoing Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-153
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Fluid Responsiveness
Keywords: the pressure gradient for venous return; fluid responsiveness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fluid infusion — 250 ml of liquid will be given within 10 minutes for each patients, and the hemodynamic parameters before and after fluid infusion will be recorded. Then the experiment is completed.

SUMMARY:
Surgical patients, especially those with insufficient blood volume and hypotension, often need fluid therapy. However, there is still a lack of simple and reliable indicators for judging transfusion responsiveness in some types of surgery. Previous studies have shown that Pressure Gradient for Venous Return (PVR) can be used to guide infusion. Thus, our aim is to explore the relationship between PVR and liquid reactivity.

DETAILED DESCRIPTION:
Fluid resuscitation is one of the key issues in the management of surgery and anesthesia. Fluid infusion test is a method to determine patients' reactivity to liquid therapy. The commonly used Stroke Volume Variation (SVV) and Pulse Pressure Variation (PPV) are good predictors of fluid responsiveness, but they are not suitable for operations with increased intra-abdominal pressure, such as laparoscopy surgery. Some studies have shown that Pressure Gradient for Venous Return (PVR) may has the same effect as PPV/SVV in predicting fluid responsiveness (FR). In the case that PPV/SVV cannot be used, PVR may be used alternatively. Therefore, our aim is to explore the relationship between the changes of PVR and fluid responsiveness during liquid infusion and to determine relevant parameters.

We will choose patients planed to receive laparoscopic surgery and general anesthesia, especially the patients with gastrointestinal tumors because of generally long operation time and much infusion volume. In our hospital, these patients will routinely indwelled arterial catheters and deep venous catheters during the operation. The former is mainly used to monitor direct arterial pressure, and the latter is used for fluid infusion.Through the above two pathways, we can collect the hemodynamic parameters of patients, and then establish the relationship between PVR and FR.

In our study, a good FR was defined as a 10% increase in cardiac index (CI) after fluid infusion, and PVR is calculated by a special formula based on some specific parameters of hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic surgery and general anesthesia

Exclusion Criteria:

* cardiac insufficiency; severe arrhythmias; patients using intra-aortic balloon pump; use of left ventricular assist devices; spasm of peripheral arteries caused by some factor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic surgery and general anesthesia
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
hemodynamic parameters | At enrollment
  direct arterial pressure including systolic, diastolic and mean arterial pressure; central venous pressure.These data are collected continuously and dynamically.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Min, Doctor, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided